CLINICAL TRIAL: NCT00812955
Title: An 8-Week, Multicenter, Randomized, Double-blind, Four-arm, Parallel-group Study Comparing the Safety and Efficacy of ABT-143 to Simvastatin in Subjects With Hypercholesterolemia
Brief Title: Safety and Efficacy Study Comparing ABT-143 to Simvastatin in Subjects With Elevated Levels of Low Density Lipoprotein Cholesterol ("Bad Cholesterol") and Triglycerides
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M10-667
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Results first posted 2012-08-01 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-09

CONDITIONS: Dyslipidemia, Hypercholesterolemia, Hypertriglyceridemia
Keywords: Dyslipidemia; Hypercholesterolemia; Hypertriglyceridemia
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia; Hypertriglyceridemia | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A - ABT-143 capsules 5/135 mg (Experimental): ABT-143 capsules 5/135 mg - ABT-143 (rosuvastatin 5 mg in combination with fenofibric acid 135 mg) once daily for 8 weeks
  Interventions: Drug: ABT-143
- B - ABT-143 capsules 10/135 mg (Experimental): ABT-143 capsules 10/135 mg - ABT-143 (rosuvastatin 10 mg in combination with fenofibric acid 135 mg) once daily for 8 weeks
  Interventions: Drug: ABT-143
- C - ABT-143 capsules 20/135 mg (Experimental): ABT-143 capsules 20/135 mg - ABT-143 (rosuvastatin 20 mg in combination with fenofibric acid 135 mg) once daily for 8 weeks
  Interventions: Drug: ABT-143
- D - Simvastatin capsules 40 mg (Active Comparator): Simvastatin capsules 40 mg daily for 8 weeks
  Interventions: Drug: simvastatin

INTERVENTIONS:
Drug: ABT-143 — Once daily for 8 weeks
  Arms: A - ABT-143 capsules 5/135 mg; B - ABT-143 capsules 10/135 mg; C - ABT-143 capsules 20/135 mg
Drug: simvastatin — Once daily for 8 weeks simvastatin capsules 40 mg
  Arms: D - Simvastatin capsules 40 mg

SUMMARY:
The primary purpose of this study is to test the effect and safety of three different doses of ABT-143 compared to simvastatin in subjects with elevated levels of low density lipoprotein cholesterol ("bad cholesterol") and triglycerides.

DETAILED DESCRIPTION:
There are 4 treatment groups in the study: ABT-143 capsules 20/135 mg, ABT-143 capsules 10/135 mg, ABT-143 5/135 mg, and simvastatin capsules 40 mg. The primary outcome measure only compares 2 of these groups: ABT-143 capsules 20/135 mg and the simvastatin capsules 40 mg groups, therefore there are only results for these 2 groups and not all 4 groups for this outcome measure . Secondary outcome measure (mean percent change in LDL-C comparing ABT-143 capsules 10/135 mg to simvastatin capsules 40 mg) only compares these 2 groups: ABT-143 capsules 10/135 mg and simvastatin capsules 40 mg, therefore there are only results for these 2 groups and not all 4 groups for this outcome measure. Secondary outcome measure (mean percent change in LDL-C comparing ABT-143 capsules 5/135 mg to simvastatin capsules 40 mg) only compares these 2 groups: ABT-143 capsules 5/135 mg and simvastatin capsules 40 mg, therefore there are only results for these 2 groups and not all 4 groups for this outcome measure. For the other pre-specified outcome measures, median percent change in triglycerides from baseline to the final visit and mean percent change in HDL-C from baseline to the final visit for the full analysis sets, all 3 ABT-143 capsules 20/135 mg, 10/135 mg, and 5/135 mg groups were compared to the simvastatin capsules 40 mg group, therefore there are results for all 4 treatment groups for these outcome measures.

ELIGIBILITY:
Inclusion Criteria

* Participants with hypercholesterolemia and hypertriglyceridemia.
* Participants had the following fasting lipid results following a greater than or equal to 12 hour fasting period (measured at the Screening Visit(s)):

  * Triglycerides level greater than or equal to 150 milligrams/deciliter (mg/dL) and less than 400 milligrams/deciliter, and
  * Low-density lipoprotein cholesterol greater than or equal to 160 milligrams/deciliter and less than or equal to 240 milligrams/deciliter.

Exclusion Criteria

* Participants with certain chronic or unstable medical conditions.
* Participants receiving coumarin anticoagulants, systemic cyclosporins, or certain other medications.
* Pregnant or lactating women, or women intending to become pregnant.
* Participants with diabetes mellitus that is poorly controlled.
* Participant was of Asian ancestry (having Filipino, Chinese, Japanese, Korean, Vietnamese, or Asian-Indian origin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Torbjörn Lundström, MD, Study Director — AstraZeneca
Locations (129):
- United States (129):
  - Site Reference ID/Investigator# 12654, Birmingham, Alabama
  - Site Reference ID/Investigator# 12634, Columbiana, Alabama
  - Site Reference ID/Investigator# 12559, Huntsville, Alabama
  - Site Reference ID/Investigator# 12499, Ozark, Alabama
  - Site Reference ID/Investigator# 12673, Chandler, Arizona
  - Site Reference ID/Investigator# 17282, Scottsdale, Arizona
  - Site Reference ID/Investigator# 12657, Little Rock, Arkansas
  - Site Reference ID/Investigator# 12489, Anaheim, California
  - Site Reference ID/Investigator# 12495, Carmichael, California
  - Site Reference ID/Investigator# 12467, Chula Vista, California
  - Site Reference ID/Investigator# 12498, Long Beach, California
  - Site Reference ID/Investigator# 12602, Los Angeles, California
  - Site Reference ID/Investigator# 12510, Norwalk, California
  - Site Reference ID/Investigator# 12550, Palm Desert, California
  - Site Reference ID/Investigator# 16503, Roseville, California
  - Site Reference ID/Investigator# 12678, Sacramento, California
  - Site Reference ID/Investigator# 14241, Sacramento, California
  - Site Reference ID/Investigator# 12473, San Diego, California
  - Site Reference ID/Investigator# 12497, Walnut Creek, California
  - Site Reference ID/Investigator# 12680, West Hills, California
  - Site Reference ID/Investigator# 12461, Colorado Springs, Colorado
  - Site Reference ID/Investigator# 12600, Colorado Springs, Colorado
  - Site Reference ID/Investigator# 12679, Waterbury, Connecticut
  - Site Reference ID/Investigator# 12598, Clearwater, Florida
  - Site Reference ID/Investigator# 15542, Coral Gables, Florida
  - Site Reference ID/Investigator# 12477, Daytona Beach, Florida
  - Site Reference ID/Investigator# 12668, Delray Beach, Florida
  - Site Reference ID/Investigator# 15483, Fort Lauderdale, Florida
  - Site Reference ID/Investigator# 12645, Fort Myers, Florida
  - Site Reference ID/Investigator# 12672, Hollywood, Florida
  - Site Reference ID/Investigator# 17504, Jacksonville, Florida
  - Site Reference ID/Investigator# 12781, Jacksonville, Florida
  - Site Reference ID/Investigator# 12665, Jupiter, Florida
  - Site Reference ID/Investigator# 12682, Longwood, Florida
  - Site Reference ID/Investigator# 15486, Melbourne, Florida
  - Site Reference ID/Investigator# 12502, New Port Richey, Florida
  - Site Reference ID/Investigator# 12647, Ocala, Florida
  - Site Reference ID/Investigator# 12520, Orlando, Florida
  - Site Reference ID/Investigator# 12687, Ormond Beach, Florida
  - Site Reference ID/Investigator# 12583, Sarasota, Florida
  - Site Reference ID/Investigator# 12652, Tampa, Florida
  - Site Reference ID/Investigator# 12557, West Palm Beach, Florida
  - Site Reference ID/Investigator# 12621, Winter Haven, Florida
  - Site Reference ID/Investigator# 16505, Winter Park, Florida
  - Site Reference ID/Investigator# 12675, Augusta, Georgia
  - Site Reference ID/Investigator# 12620, Dunwoody, Georgia
  - Site Reference ID/Investigator# 12653, Roswell, Georgia
  - Site Reference ID/Investigator# 12555, Suwanee, Georgia
  - Site Reference ID/Investigator# 12787, Woodstock, Georgia
  - Site Reference ID/Investigator# 12514, Chicago, Illinois
  - Site Reference ID/Investigator# 12487, Peoria, Illinois
  - Site Reference ID/Investigator# 12627, Peoria, Illinois
  - Site Reference ID/Investigator# 12529, Evansville, Indiana
  - Site Reference ID/Investigator# 12688, Indianapolis, Indiana
  - Site Reference ID/Investigator# 15485, South Bend, Indiana
  - Site Reference ID/Investigator# 12676, Arkansas City, Kansas
  - Site Reference ID/Investigator# 12597, Wichita, Kansas
  - Site Reference ID/Investigator# 12472, Louisville, Kentucky
  - Site Reference ID/Investigator# 12658, Mount Sterling, Kentucky
  - Site Reference ID/Investigator# 12586, Baltimore, Maryland
  - Site Reference ID/Investigator# 12480, Bethesda, Maryland
  - Site Reference ID/Investigator# 12638, Oxon Hill, Maryland
  - Site Reference ID/Investigator# 12513, Springfield, Massachusetts
  - Site Reference ID/Investigator# 12663, Kalamazoo, Michigan
  - Site Reference ID/Investigator# 12609, Brooklyn Center, Minnesota
  - Site Reference ID/Investigator# 16622, Edina, Minnesota
  - Site Reference ID/Investigator# 12625, Jackson, Mississippi
  - Site Reference ID/Investigator# 12560, Olive Branch, Mississippi
  - Site Reference ID/Investigator# 12534, City of Saint Peters, Missouri
  - Site Reference ID/Investigator# 12677, St Louis, Missouri
  - Site Reference ID/Investigator# 12592, Billings, Montana
  - Site Reference ID/Investigator# 12655, Omaha, Nebraska
  - Site Reference ID/Investigator# 12587, Las Vegas, Nevada
  - Site Reference ID/Investigator# 12554, Berlin, New Jersey
  - Site Reference ID/Investigator# 12637, Elizabeth, New Jersey
  - Site Reference ID/Investigator# 12463, Hillsborough, New Jersey
  - Site Reference ID/Investigator# 12660, Trenton, New Jersey
  - Site Reference ID/Investigator# 12506, Albuquerque, New Mexico
  - Site Reference ID/Investigator# 12539, Johnson City, New York
  - Site Reference ID/Investigator# 12631, Syracuse, New York
  - Site Reference ID/Investigator# 17503, Cary, North Carolina
  - Site Reference ID/Investigator# 12650, Charlotte, North Carolina
  - Site Reference ID/Investigator# 12504, Charlotte, North Carolina
  - Site Reference ID/Investigator# 12558, Charlotte, North Carolina
  - Site Reference ID/Investigator# 12671, Charlotte, North Carolina
  - Site Reference ID/Investigator# 12527, Hickory, North Carolina
  - Site Reference ID/Investigator# 12608, Morehead City, North Carolina
  - Site Reference ID/Investigator# 12535, Salisbury, North Carolina
  - Site Reference ID/Investigator# 12656, Statesville, North Carolina
  - Site Reference ID/Investigator# 17641, Wilmington, North Carolina
  - Site Reference ID/Investigator# 12606, Winston-Salem, North Carolina
  - Site Reference ID/Investigator# 12614, Akron, Ohio
  - Site Reference ID/Investigator# 12662, Cincinnati, Ohio
  - Site Reference ID/Investigator# 12545, Cincinnati, Ohio
  - Site Reference ID/Investigator# 12640, Kettering, Ohio
  - Site Reference ID/Investigator# 12786, Mason, Ohio
  - Site Reference ID/Investigator# 12630, Warren, Ohio
  - Site Reference ID/Investigator# 12551, Oklahoma City, Oklahoma
  - Site Reference ID/Investigator# 12611, Tulsa, Oklahoma
  - Site Reference ID/Investigator# 12585, Medford, Oregon
  - Site Reference ID/Investigator# 12610, Beaver, Pennsylvania
  - Site Reference ID/Investigator# 12589, Duncansville, Pennsylvania
  - Site Reference ID/Investigator# 12607, Harleysville, Pennsylvania
  - Site Reference ID/Investigator# 12641, Jersey Shore, Pennsylvania
  - Site Reference ID/Investigator# 12507, Melrose Park, Pennsylvania
  - Site Reference ID/Investigator# 12624, Perkasie, Pennsylvania
  - Site Reference ID/Investigator# 12669, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 12788, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 12525, Pittsburgh, Pennsylvania
  - Site Reference ID/Investigator# 12601, Tipton, Pennsylvania
  - Site Reference ID/Investigator# 12686, Warminster, Pennsylvania
  - Site Reference ID/Investigator# 12623, Mt. Pleasant, South Carolina
  - Site Reference ID/Investigator# 12681, Mt. Pleasant, South Carolina
  - Site Reference ID/Investigator# 12485, Simpsonville, South Carolina
  - Site Reference ID/Investigator# 12639, Summerville, South Carolina
  - Site Reference ID/Investigator# 15642, Germantown, Tennessee
  - Site Reference ID/Investigator# 12643, Jackson, Tennessee
  - Site Reference ID/Investigator# 12470, Dallas, Texas
  - Site Reference ID/Investigator# 16081, Dallas, Texas
  - Site Reference ID/Investigator# 12492, Dallas, Texas
  - Site Reference ID/Investigator# 12464, Fort Worth, Texas
  - Site Reference ID/Investigator# 12646, San Antonio, Texas
  - Site Reference ID/Investigator# 16601, San Antonio, Texas
  - Site Reference ID/Investigator# 12540, San Antonio, Texas
  - Site Reference ID/Investigator# 12466, San Antonio, Texas
  - Site Reference ID/Investigator# 12622, San Antonio, Texas
  - Site Reference ID/Investigator# 12538, Norfolk, Virginia
  - Site Reference ID/Investigator# 12616, Richmond, Virginia
  - Site Reference ID/Investigator# 12476, Madison, Wisconsin

REFERENCES:
- [Derived] Roth EM, McKenney JM, Kelly MT, Setze CM, Carlson DM, Gold A, Stolzenbach JC, Williams LA, Jones PH. Efficacy and safety of rosuvastatin and fenofibric acid combination therapy versus simvastatin monotherapy in patients with hypercholesterolemia and hypertriglyceridemia: a randomized, double-blind study. Am J Cardiovasc Drugs. 2010;10(3):175-86. doi: 10.2165/11533430-000000000-00000. PMID 20524719

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 474 subjects were randomized and treated at 111 sites in the United States between 29 December 2008 and 14 May 2009.
Groups:
- Simvastatin Capsules 40 mg: Simvastatin capsules 40 mg once daily for 8 weeks
- ABT-143 Capsules 5/135 mg: ABT-143 capsules 5/135 mg once daily for 8 weeks
- ABT-143 Capsules 10/135 mg: ABT-143 capsules 10/135 mg once daily for 8 weeks
- ABT-143 Capsules 20/135 mg: ABT-143 capsules 20/135 mg once daily for 8 weeks
Period: Overall Study
Arm/Group | Simvastatin Capsules 40 mg | ABT-143 Capsules 5/135 mg | ABT-143 Capsules 10/135 mg | ABT-143 Capsules 20/135 mg
Started | 119 | 118 | 119 | 118
Completed | 109 | 111 | 113 | 110
Not Completed | 10 | 7 | 6 | 8
Not completed — Adverse Event | 7 | 6 | 3 | 4
Not completed — Lost to Follow-up | 2 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 2
Not completed — randomized in error | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin Capsules 40 mg | ABT-143 Capsules 5/135 mg | ABT-143 Capsules 10/135 mg | ABT-143 Capsules 20/135 mg | Total
Number analyzed (Participants) | 119 | 118 | 119 | 118 | 474
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 92 | 91 | 95 | 95 | 373
  >=65 years | 27 | 27 | 24 | 23 | 101
Age Continuous [Mean (Standard Deviation); unit: years] | 56.8 (9.77) | 56.8 (8.91) | 56.6 (9.27) | 56.0 (10.41) | 56.6 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 62 | 59 | 60 | 252
  Male | 48 | 56 | 60 | 58 | 222
Region of Enrollment [Number; unit: participants]
  United States | 119 | 118 | 119 | 118 | 474

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline to the Final Visit in Low-density Lipoprotein Cholesterol (LDL-C) (Full Analysis Set)
Description: The mean percent change from Baseline to the Final Visit in low-density lipoprotein cholesterol, comparing the following two treatment groups:
  ABT-143 capsules 20/135 milligrams versus simvastatin capsules 40 milligrams for the full analysis set.
Time Frame: Baseline to 8 weeks
Population: Full Analysis Set was used and defined as all randomized participants who had both a baseline value and at least 1 post-baseline value for LDL-C. Last observation carried forward (LOCF) was used to impute values for participants missing a post-baseline visit value. Only post-baseline values were carried forward.
Measure: Mean (Standard Error); unit: percent change
Groups:
- Simvastatin Capsules 40 mg: Simvastatin capsules 40 mg
- ABT-143 Capsules 20/135 mg: ABT-143 capsules 20/135 mg
Arm/Group | Simvastatin Capsules 40 mg | ABT-143 Capsules 20/135 mg
Number analyzed (Participants) | 114 | 113
percent change | -32.8 (1.59) | -47.2 (1.60)

2. Secondary Outcome: Mean Percent Change From Baseline to the Final Visit in Low-density Lipoprotein Cholesterol (LDL-C), With ABT-143 Capsules 10/135 Milligrams Versus Simvastatin Capsules 40 Milligrams (Full Analysis Set)
Description: The mean percent change from Baseline to the Final Visit in low-density lipoprotein cholesterol, comparing the following treatment groups, ABT-143 capsules 10/135 milligrams versus simvastatin capsules 40 milligrams for the full analysis set.
Time Frame: Baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percent change
Groups:
- ABT-143 Capsules 10/135 mg: ABT-143 capsules 10/135 mg
Arm/Group | Simvastatin Capsules 40 mg | ABT-143 Capsules 10/135 mg
Number analyzed (Participants) | 114 | 115
percent change | -32.8 (1.59) | -46.0 (1.59)

3. Secondary Outcome: Mean Percent Change From Baseline to the Final Visit in Low-density Lipoprotein Cholesterol (LDL-C), With ABT-143 Capsules 5/135 Milligrams Versus Simvastatin Capsules 40 Milligrams (Full Analysis Set)
Description: The mean percent change from Baseline to the Final Visit in low-density lipoprotein cholesterol, comparing the following treatment groups, ABT-143 capsules 5/135 milligrams versus simvastatin capsules 40 milligrams for the full analysis set.
Time Frame: Baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percent change
Groups:
- ABT-143 Capsules 5/135 mg: ABT-143 capsules 5/135 mg
Arm/Group | Simvastatin Capsules 40 mg | ABT-143 Capsules 5/135 mg
Number analyzed (Participants) | 114 | 114
percent change | -32.8 (1.59) | -38.9 (1.59)

4. Other Pre Specified Outcome: Median Percent Change in Triglycerides From Baseline to the Final Visit (Full Analysis Set)
Description: The ABT-143 capsules 20/135 milligram, ABT-143 capsules 10/135 milligram, and ABT-143 capsules 5/135 milligram groups were compared to the simvastatin capsules 40 milligram group for median percent change in triglycerides from Baseline to the Final Visit for the full analysis set.
Time Frame: Baseline to 8 weeks
Population: Full Analysis Set was used and defined as all randomized participants who had both a baseline value and at least 1 post-baseline value for triglycerides. Last observation carried forward (LOCF) was used to impute values for participants missing a post-baseline visit value. Only post-baseline values were carried forward.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Simvastatin Capsules 40 mg | ABT-143 Capsules 5/135 mg | ABT-143 Capsules 10/135 mg | ABT-143 Capsules 20/135 mg
Number analyzed (Participants) | 114 | 114 | 115 | 113
percent change | -20.8 [-41.3 to 1.9] | -42.7 [-54.5 to -30.4] | -44.6 [-55.4 to -31.6] | -50.0 [-57.5 to -32.1]

5. Other Pre Specified Outcome: Mean Percent Change in High-density Lipoprotein Cholesterol (HDL-C) From Baseline to the Final Visit (Full Analysis Set)
Description: The ABT-143 capsules 20/135 milligram, ABT-143 capsules 10/135 milligram, and ABT-143 capsules 5/135 milligram groups were compared to the simvastatin capsules 40 milligram group for mean percent change in high-density lipoprotein cholesterol from Baseline to the Final Visit for the full analysis set.
Time Frame: Baseline to 8 weeks
Population: Full Analysis Set was used and defined as all randomized participants who had both a baseline value and at least 1 post-baseline value for HDL-C. Last observation carried forward (LOCF) was used to impute values for participants missing a post-baseline visit value. Only post-baseline values were carried forward.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Simvastatin Capsules 40 mg | ABT-143 Capsules 5/135 mg | ABT-143 Capsules 10/135 mg | ABT-143 Capsules 20/135 mg
Number analyzed (Participants) | 114 | 114 | 115 | 113
percent change | 9.6 (1.56) | 16.2 (1.56) | 14.0 (1.55) | 15.7 (1.56)

ADVERSE EVENTS:
Time Frame: 18 weeks
Description: Treatment-emergent adverse events were defined as those occurring after study drug initiation and within 30 days after the last dose of study drug. Serious adverse events were collected from the time the participant signed the informed consent until 30 calendar days following discontinuation of study drug.
Arm/Group | Simvastatin Capsules 40 mg | ABT-143 Capsules 5/135 mg | ABT-143 Capsules 10/135 mg | ABT-143 Capsules 20/135 mg
Serious Adverse Events (participants affected / at risk) | 0/119 | 4/118 | 1/119 | 3/118
Other Adverse Events (participants affected / at risk) | 10/119 | 13/118 | 6/119 | 17/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Simvastatin Capsules 40 mg (N=119) | ABT-143 Capsules 5/135 mg (N=118) | ABT-143 Capsules 10/135 mg (N=119) | ABT-143 Capsules 20/135 mg (N=118)
Angina Pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Abdominal Hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 0 | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Simvastatin Capsules 40 mg (N=119) | ABT-143 Capsules 5/135 mg (N=118) | ABT-143 Capsules 10/135 mg (N=119) | ABT-143 Capsules 20/135 mg (N=118)
Nausea (Gastrointestinal disorders) | 2 | 7 | 3 | 6
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 2 | 2 | 7
Headache (Nervous system disorders) | 8 | 5 | 1 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.